CLINICAL TRIAL: NCT04421092
Title: Efficacy of Superior Laryngeal Nerve Block for Chronic Cough
Brief Title: Efficacy of SLN Block for Chronic Cough
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 00096384
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Results first posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-09

CONDITIONS: Cough; Superior Laryngeal Nerve Block; Neurogenic Cough
Keywords: superior laryngeal nerve block; chronic cough
MeSH Terms: conditions — Cough; Chronic Cough | interventions — Sodium Chloride; Triamcinolone; Lidocaine; Epinephrine

STUDY DESIGN:
Intervention Model Description: Two treatment arms:
  1. Treatment Group (n=25) - 2 mL of 1:1 triamcinolone 40:1% lidocaine with 1:2000000 epinephrine.
  2. Placebo group (n=25) 2 mL of saline.
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Steroid-Lidocaine Mixture (Experimental): Will receive numbing injection, which is a mixture of steroid and lidocaine
  Interventions: Procedure: Superior laryngeal nerve block; Procedure: Injection of steroid-lidocaine mixture
- Placebo (Placebo Comparator): Will receive saline injection as a placebo
  Interventions: Procedure: Superior laryngeal nerve block; Procedure: Injection of placebo (saline)

INTERVENTIONS:
Procedure: Superior laryngeal nerve block — Injection of either the steroid-lidocaine mixture or placebo through the skin around where the superior laryngeal nerve is located on the neck. The procedure lasts 5 minutes and is done in the clinic.
  Other Names: Injection of steroid-lidocaine mixture vs. placebo (saline)
Procedure: Injection of placebo (saline) — Superior laryngeal nerve block using 1mL of saline as the injection.
  Other Names: 1mL of saline as the injection
  Arms: Placebo
Procedure: Injection of steroid-lidocaine mixture — Superior laryngeal nerve block using 1mg 1:1 triamcinolone 40mg: 1% lidocaine with 1:200000 epinephrine as the injection.
  Other Names: 1mg 1:1 triamcinolone 40mg: 1% lidocaine with 1:200000 epinephrine as the injection.
  Arms: Steroid-Lidocaine Mixture

SUMMARY:
This is a research study to find out if superior laryngeal nerve blocks are an effective way to reduce cough when compared to placebo (a substance without any medical value). Eligibility for the study include the following: age >18, cough history suggestive that the nerve to the voice box is overactive, non-smoker, Patients will be followed over time and assigned to either the treatment or placebo group at random. The treatment would be four superior laryngeal nerve blocks and the placebo would be four saline injections (the inactive substance). Study team will measure if the injection improved cough and ask patients to keep a log of symptoms and fill out questionnaires at each visit. After the four injections, patients will follow up in 3 months to see if cough has returned and if so, how severe the cough is.

ELIGIBILITY:
Inclusion Criteria:

* History consistent with neurogenic cough
* Exclusion of other etiologies (see exclusion criteria)
* Age ≥ 18

Exclusion Criteria:

* Current neuromodulating medication use
* Untreated other etiologies of cough:

Current smoker Current ACE/ARB use Abnormal PFTs within 6 months Uncontrolled OSA Abnormal CXR within 6 months RSI > 13 or RFS >11 AND workup positive for GERD (esophagram, 24-hour pH probe, manometry, EGD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Tipton, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects will be recruited within the standard workup for chronic cough in the clinic. Patients will be screened at the initial visit if they meet inclusion criteria or at further visits after additional workup for other sources of cough is completed, patients will be offered participation in the study. The principal investigator will discuss risks and benefits of study participation with the eligible subjects using the informed consent form.
Period: Overall Study
Arm/Group | Steroid-Lidocaine Mixture | Placebo
Started (10) | 7 | 10
Completed | 7 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: LCQ scores, VAS scores
Groups:
- Total: Total of all reporting groups
Arm/Group | Steroid-Lidocaine Mixture | Placebo | Total
Number analyzed (Participants) | 10 | 7 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 7 | 17
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 56.3 [18 to 65] | 56.3 [18 to 65] | 56.3 [18 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 8 | 7 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Change in Cough Severity
Description: Patient will complete the Leicester Cough Questionnaire at each visit. This is a validated survey that measures 3 domains (physical, psychological and social). The total score range is 3-21 and domain scores range from 1-7; a higher score indicates a better quality of life.
Time Frame: Change from Baseline to 3 months
Measure: Mean (Standard Deviation); unit: LCQ scores (baseline to 3 months)
Arm/Group | Steroid-Lidocaine Mixture | Placebo
Number analyzed (Participants) | 10 | 7
LCQ scores (baseline to 3 months) | 13.15 (4.52) | 9.54 (3.87)

2. Secondary Outcome: Subjective Improvement in Cough
Description: Improvement was defined as a 'yes' response at any time point during the study (1-4 weeks or 3 months post-treatment). The reported value reflects the total number of participants who reported improvement at any time point.
Time Frame: Baseline, 1-4 weeks post-injection, and 3 months post-treatment
Measure: Number; unit: participants
Arm/Group | Steroid-Lidocaine Mixture | Placebo
Number analyzed (Participants) | 10 | 7
participants | 10 | 7

3. Secondary Outcome: Summed Daily Change in Subjective Cough Severity
Description: Participants rate cough severity on a 0-15 visual analogue scale. Scores are recorded daily and analyzed using regression. Higher scores indicate greater severity. VAS is a 0-15 scale completed daily by participants.
  Severity is measured using a ruler to determine percentage along the scale. Scores were analyzed using regression models to assess trends over time.
Time Frame: Daily for 3 months post-injection
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid-Lidocaine Mixture | Placebo
Number analyzed (Participants) | 10 | 7
score on a scale | 13.15 (4.52) | 9.54 (3.87)

ADVERSE EVENTS:
Time Frame: 1 year and 6 months
Description: This is a routine procedure done by laryngologists.
Arm/Group | Steroid-Lidocaine Mixture | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/7
Other Adverse Events (participants affected / at risk) | 3/10 | 1/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Steroid-Lidocaine Mixture (N=10) | Placebo (N=7)
Mild transient soreness at injection site (Investigations) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-20): https://cdn.clinicaltrials.gov/large-docs/92/NCT04421092/Prot_SAP_000.pdf